CLINICAL TRIAL: NCT02704195
Title: Subthalamic Nucleus Stimulation Effect on Gait Symmetry and Freezing of Gait
Acronym: STIMSYM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-A01323-42
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Deep brain stimulation; Freezing of Gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic Subthalamic nucleus stimulation (Active Comparator): This arm is the reference, with the best stimulation parameters
  Interventions: Procedure: Chronic Subthalamic nucleus stimulation
- Unilateral reduction of stimulation (Experimental): 30% unilateral reduction of Subthalamic nucleus stimulation
  Interventions: Procedure: Unilateral reduction of stimulation

INTERVENTIONS:
Procedure: Unilateral reduction of stimulation — 30% unilateral reduction of Subthalamic nucleus stimulation
  Arms: Unilateral reduction of stimulation
Procedure: Chronic Subthalamic nucleus stimulation — This arm is the reference, with the best stimulation parameters
  Arms: Chronic Subthalamic nucleus stimulation

SUMMARY:
Impact of unilateral modulation of deep brain stimulation of the subthalamic nucleus on freezing of gait in Parkinson's disease

DETAILED DESCRIPTION:
Unilateral modulation of subthalamic stimulation and its impact on freezing of gait in Parkinson's disease will be studied.

In a cross-over, doubleblind, randomized study, a 30% reduction of stimulation intensity of the less impacted side will be compared with chronic treatment with regard to frequency and duration of freezing of gait episodes.

ELIGIBILITY:
Inclusion Criteria:

Patients affiliated to social security Patient with idiopathic parkinson's disease, with deep brain stimulation since at least one year Freezing of gait Able to give inform consent

Exclusion Criteria:

Patient under guardianship, legal guardianship Psychosis Severe depression Severe cognitive troubles (Mattis < 130) Other neurologic or medical pathology interfering with gait

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
improvement of Freezing of gait | 1 month after new stimulation parameters
  the improvement will be measure with a composite score of items 12 + 13 on UPDRS II and items 10+11 on UPDRS III,

CONTACTS AND LOCATIONS:
Overall Officials: Elena Moro, MD, Study Director — University Hospital, Grenoble
Locations (1):
- CHU Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meoni S, Debu B, Pelissier P, Scelzo E, Castrioto A, Seigneuret E, Chabardes S, Fraix V, Moro E. Asymmetric STN DBS for FOG in Parkinson's disease: A pilot trial. Parkinsonism Relat Disord. 2019 Jun;63:94-99. doi: 10.1016/j.parkreldis.2019.02.032. Epub 2019 Feb 25. PMID 30826266